CLINICAL TRIAL: NCT01987804
Title: A Double-blind, Placebo Controlled Single Centre Trial to Evaluate the Dose-relationship of the Effects of Vaginally Administered Oxytocin on the Vaginal Mucosal Membrane in Postmenopausal Women With Vaginal Atrophy
Brief Title: Dose-relationship of Vaginally Administrated Oxytocin in Postmenopausal Women
Acronym: OXYPEP002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXYPEP002
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin 100 i.u. (Experimental): N=24 patients are administrated Oxytocin 100 i.u. vaginally
  Interventions: Drug: Oxytocin 100 i.u.
- Oxytocin 400 i.u. (Experimental): N=24 patients are administrated Oxytocin 400 i.u. vaginally
  Interventions: Drug: Oxytocin 400 i.u.
- Placebo (Placebo Comparator): N=16 patients are administrated placebo vaginally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin 100 i.u.
  Other Names: Vagoticin
  Arms: Oxytocin 100 i.u.
Drug: Oxytocin 400 i.u.
  Other Names: Vagoticin
  Arms: Oxytocin 400 i.u.
Drug: Placebo
  Arms: Placebo

SUMMARY:
Up to 50% of all postmenopausal women, experience vaginal drynes, i.e. vaginal atrophy is a consequence due to the lack of estrogen. In addition, vaginal atrophy is associated with an increased pH, which creates an environment more susceptible to infections . The mucosal epithelium shows signs of severe senile atrophy and cytological examination demonstrate increased number of the basal and parabasal cells and reduced number of superficial cells . Unlike some other menopausal symptoms (for instance hot flushes), vaginal symptoms generally persist or worsen with aging.Oxytocin is a peptide hormone and it is released systemically via the posterior pituitary. The most well known effects of oxytocin are its roles in female reproduction such as facilitation of birth and breast feeding. Oxytocin has also shown to exert positive effects on the proliferation of human vaginal mucosal cells from postmenopausal women, an effect which could be attributed either to the direct stimulation of new cell formation or to an increased production of other growth factors. The primary objective is to investigate the dose relationsship of topical administrated Vagitocin on the vaginal mucosal membrane, measured in the change (%)of superficial cells up to 7 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Naturally postmenopausal or ooforectomized women, completely without menstrual bleedings for at least four years prior to baseline.
2. > 40 years of age.
3. Moderate to severe symptoms of at least one of the following criteria of vulvar and vaginal atrophy associated with the menopause, according to the patient's self-assessement: vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity, or presence of vaginal bleeding associated with sexual activity.
4. Atrophic mucosa according to the investigator's assessment.
5. Signed Informed Consent.

Exclusion Criteria:

* 1. Usage of any sex steroids including phytoestrogens, hormonal intra-uterine device or herbal medicinal products with known estrogenic effects within 3 months prior to baseline.

  2. Usage of any lubricant for intra-vaginal administration at baseline. 3. Vaginal bleeding of unknown origin. 4. Vaginal pH ≤ 5.0. 5. Any ongoing uro-genital infection within 7 days prior to baseline. 6. Body Mass Index (BMI) >30 kg/m2. 7. Systolic Blood Pressure > 150 mmHg and Diastolic Blood Pressure > 90 mmHg at baseline.

  8. Any concurrent known or suspected tumor disease as judged by the investigator.

  9. Clinically significant medical history (excluding medically well-controlled hypertension and hypercholesterolemia), abnormal findings from physical examinations, vital signs, cytology, histology, US examination of uterus and ovaries or laboratory analyses that may interfere with the trial objectives or compromise the safety of the patient as judged by the Investigator.

  10. Concurrent and diagnosed nephrological or hepatic disorder 11. Diagnosed with HIV, Hepatitis B or C 12. Known or suspected drug or alcohol abuse, within 12 months prior to baseline.

  13. Known or suspected allergy to any ingredient of the trial product. 14. Incapacity to perform trial procedures, as judged by the investigator. 15. Participation in any other interventional clinical trial within 3 months prior to baseline.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To investigate the dose-relationship of topical Vagitocin on the vaginal mucosal membrane. | from baseline visit to 7 weeks of treatment
  Change in percentage points of superficial cells from baseline visit (visit 1) to 7 weeks of treatment (Visit 3).

SECONDARY OUTCOMES:
To investigate the safety and tolerability of topical Vagitocin treatment. | From visit 2 to visit 7
  Change in percentage points of superficial cells from baseline visit to 2 (Visit 2) weeks of treatment.
  Change in maturation value from baseline visit to 2 (Visit 2) and 7 (Visit 3) weeks of treatment.
  Change in vaginal pH from baseline visit to 2 (Visit 2) and 7 (Visit 3) weeks of treatment.
  Visual appearance of the vaginal mucosa after 2 (Visit 2) and 7 (Visit 3) weeks of treatment
  * Patients´ self-assessment of the most bothersome symptomafter 2 (Visit 2), 7 (Visit 3), weeks of treatment and at the telephone follow-up after 9 weeks.
  * Histological assessment after 2 (Visit 2) and 7 weeks (Visit 3) of treatment.
  * Change in score in selected items of WHQ/SSP from baseline visit to 7 (Visit 3) weeks of treatment and at the telephone follow-up after 9 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Aino F Jonasson, M.D, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Huddinge, Sweden